CLINICAL TRIAL: NCT05762874
Title: Safety and Effectiveness of Ruxolitinib in Patients With Myelofibrosis
Brief Title: Ruxolitinib in Patients With Myelofibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ali Mahmoud Hassan, principle investigator, Assiut University
Other Study IDs: myelofibrosis
Record Dates: First submitted 2023-02-11; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Ruxolitinib — JAK inhibitor

SUMMARY:
Prospective study to evaluate the response of myelofibrosis patients to ruxolitinib and it's adverse events on patients (1 year observational study).

DETAILED DESCRIPTION:
Myelofibrosis (MF) is a clonal disorder of the pluripotent hematopoietic stem cell in which the abnormal stem cell population releases several cytokines and growth factors into the bone marrow microenvironment, it is pathologically characterized by bone marrow fibrosis, extramedullary hematopoiesis, and an overactive Janus kinase/signal transducers and activators of transcription( JAK-STAT) pathway, MF is estimated to have an annual incidence of 0.47-1.98 per 100,000, Most patients are aged > 60 years at initial diagnosis tends to be more common in males than females, It may be de novo (primary MF) or secondary to polycythemia vera (PV) or essential thrombocythemia (ET).

Most patients present with anemia, splenomegaly, and constitutional symptoms, but up to 30% of patients are asymptomatic at diagnosis, symptomatic patients develop Splenomegaly-related symptoms such as abdominal distension and pain, early satiety, dyspnea, together with constitutional symptoms such as fatigue, night sweats, cachexia, pruritus, bone pain, weight loss, and fever are the dominant aspects of the clinical picture heavily affecting the functional status and quality of life (QoL) of MF patients, the most frequent cause of death is the evolution to acute myeloid leukemia, also other conditions such as progression without transformation, cytopenia-related complications and cardiovascular events may be fatal.

Approximately 90% of patients with MF carry mutations in any of 3 driver genes: Janus kinase 2 (JAK2) in ~ 60% of cases, calreticulin (CALR) in ~ 20%, and myeloproliferative leukemia virus oncogene (MPL) in ~ 10%, Mutant proteins activate the (JAK-STAT) pathway and other pathways downstream leading to myeloproliferation, proinflammatory cytokine expression, and bone marrow remodeling.

Current diagnosis of PMF is based on the 2016 WHO-criteria and involves a composite assessment of clinical and laboratory features, Prognosis is currently based on three different scoring systems (IPSS, DIPSS, DIPSS PLUS) and recently mutations were considered in the development of three new prognostic models in PMF.

At present the only curative treatment for MF is allogeneic stem cell transplantation. Most patients with MF are considered ineligible for transplantation because of age or comorbidities, so treatment for the majority of patients is focused on symptom control.

Since the discovery of the JAK2 mutations and the development of JAK inhibitors have significantly changed the therapeutic outcome of MF as far symptoms control and patients' QoL are concerned, In this article, we present our recommendations for the practical management of MF with ruxolitinib a Janus kinase (JAK1/JAK2) inhibitor approved by the European Medicines Agency for the treatment of disease-related splenomegaly or symptoms in adult patients with primary MF , post-polycythemia vera MF , and post-essential thrombocythemia MF, and by the US Food and Drug Administration for intermediate or high-risk MF, including PMF, PPV-MF, and PET-MF. ruxolitinib therapeutic effect was not limited to Spleen volume response, being also efficacious in relieving constitutional symptoms; reducing abdominal discomfort, appetite loss, itching, fatigue, night sweats; and improving QoL. The main toxicity of ruxolitinib is hematological due to the non-selective inhibition of JAK-STAT signaling, an essential pathway for normal hematopoiesis, Due to its impairing activity on immune response, ruxolitinib may favor an increased incidence of both opportunistic and non-opportunistic infections .Few studies evaluate the role of ruxolitinib in MF and it's role in improving the patient's QoL in Assiut university so we decided to perform this influential study to assess the effectiveness of ruxolitinb in MF and it's adverse events on MF patients.

ELIGIBILITY:
Inclusion Criteria:

* PMF was diagnosed according to the 2016 revised International Standard Criteria, and PPV-MF or PET-MF according to standard criteria with JAK2 positive mutation , palpable spleen (≥5 cm below the left costal margin, measured using a soft ruler during quiet respiration), high-risk and intermediate-2 risk PMF, PPV-MF or PET-MF with disease-related symptoms or symptomatic splenomegaly and patients with intermediate-1 risk PMF, PPV-MF or PET-MF who have symptoms not controlled with supportive therapies or symptomatic splenomegaly .
* patients who previously started Ruxolitinib and still taking it .

Exclusion Criteria:

* low risk MF patients
* intermediate risk 1 without splenomegaly or symptoms
* JAK2 negative mutation
* inadequate bone marrow reserve at baseline visit, as demonstrated by at least 1 of the following: absolute neutrophil count (ANC) ≤1 × 109/l, platelet count <50 × 109/l, without the assistance of growth factors, thrombopoietic factors or platelet transfusions, and Hb ≤6.5 g/dl despite transfusions
* severely impaired renal function (defined by creatinine clearance less than 30 ml/min); inadequate liver function (total bilirubin ≥2.5 × upper limit of normal [ULN] and subsequent determination of direct bilirubin ≥2.5 × ULN or alanine aminotransferase >2.5 × ULN or aspartate aminotransferase >2.5 × ULN
* acute viral hepatitis or active chronic hepatitis B or C infection
* concurrent treatment with a potent systemic inhibitor or inducer of CYP3A4

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients who are attending clinical hematology unit and clinic in Assiut university are evaluated for:
  1. diagnosis (before start of treatment for naive patients)
  2. if confirmed diagnosis (for naive and previously diagnosed patients)
  3. follow up at (3,6,12 months) by
     * CBC
     * spleen size
     * symptoms burden according to MF-SAF (symptom assessment form)
     * Transfusion demand
     * dosage adjustment, treatment duration and discontinuation rates
  4. Adverse events of the drug mainly hematological cytopenia according to WHO criteria of drug toxicity and hepatitis infection or reactivation
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
decrease of spleen size | 6 months
  the proportion of patients achieving ≥50% reduction in Spleen size
symptoms burden | 6 months
  change in the burden of the constitutional symptoms assessed by the MF Symptom Assessment Form on a scale of 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be)

SECONDARY OUTCOMES:
adverse events of Ruxolitinib on myleofibrosis patients according to WHO criteria of drug toxicity | 1 year
  Anemia,leucopenia and thrombocytopenia in complete blood count and reactivation of hepatitis (B,C) virus by PCR

REFERENCES:
- [Background] Jacobson RJ, Salo A, Fialkow PJ. Agnogenic myeloid metaplasia: a clonal proliferation of hematopoietic stem cells with secondary myelofibrosis. Blood. 1978 Feb;51(2):189-94. PMID 620081
- [Background] Barosi G. Myelofibrosis with myeloid metaplasia: diagnostic definition and prognostic classification for clinical studies and treatment guidelines. J Clin Oncol. 1999 Sep;17(9):2954-70. doi: 10.1200/JCO.1999.17.9.2954. PMID 10561375
- [Background] Tefferi A. Primary myelofibrosis: 2019 update on diagnosis, risk-stratification and management. Am J Hematol. 2018 Dec;93(12):1551-1560. doi: 10.1002/ajh.25230. Epub 2018 Oct 26. PMID 30039550
- [Background] Titmarsh GJ, Duncombe AS, McMullin MF, O'Rorke M, Mesa R, De Vocht F, Horan S, Fritschi L, Clarke M, Anderson LA. How common are myeloproliferative neoplasms? A systematic review and meta-analysis. Am J Hematol. 2014 Jun;89(6):581-7. doi: 10.1002/ajh.23690. PMID 24971434
- [Background] Moulard O, Mehta J, Fryzek J, Olivares R, Iqbal U, Mesa RA. Epidemiology of myelofibrosis, essential thrombocythemia, and polycythemia vera in the European Union. Eur J Haematol. 2014 Apr;92(4):289-97. doi: 10.1111/ejh.12256. Epub 2014 Feb 3. PMID 24372927
- [Background] Cervantes F, Dupriez B, Pereira A, Passamonti F, Reilly JT, Morra E, Vannucchi AM, Mesa RA, Demory JL, Barosi G, Rumi E, Tefferi A. New prognostic scoring system for primary myelofibrosis based on a study of the International Working Group for Myelofibrosis Research and Treatment. Blood. 2009 Mar 26;113(13):2895-901. doi: 10.1182/blood-2008-07-170449. Epub 2008 Nov 6. PMID 18988864
- [Background] Shammo JM, Stein BL. Mutations in MPNs: prognostic implications, window to biology, and impact on treatment decisions. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):552-560. doi: 10.1182/asheducation-2016.1.552. PMID 27913528
- [Background] Palandri F, Palumbo GA, Iurlo A, Polverelli N, Benevolo G, Breccia M, Abruzzese E, Tiribelli M, Bonifacio M, Tieghi A, Isidori A, Martino B, Sgherza N, D'Adda M, Bergamaschi M, Crugnola M, Cavazzini F, Bosi C, Binotto G, Auteri G, Latagliata R, Ibatici A, Scaffidi L, Penna D, Cattaneo D, Soci F, Trawinska M, Russo D, Cuneo A, Semenzato G, Di Raimondo F, Aversa F, Lemoli RM, Heidel F, Reggiani MLB, Bartoletti D, Cavo M, Catani L, Vianelli N. Differences in presenting features, outcome and prognostic models in patients with primary myelofibrosis and post-polycythemia vera and/or post-essential thrombocythemia myelofibrosis treated with ruxolitinib. New perspective of the MYSEC-PM in a large multicenter study⁎. Semin Hematol. 2018 Oct;55(4):248-255. doi: 10.1053/j.seminhematol.2018.05.013. Epub 2018 Jun 5. PMID 30502854
- [Background] Barbui T, Thiele J, Gisslinger H, Kvasnicka HM, Vannucchi AM, Guglielmelli P, Orazi A, Tefferi A. The 2016 WHO classification and diagnostic criteria for myeloproliferative neoplasms: document summary and in-depth discussion. Blood Cancer J. 2018 Feb 9;8(2):15. doi: 10.1038/s41408-018-0054-y. PMID 29426921
- [Background] Tefferi A, Guglielmelli P, Lasho TL, Gangat N, Ketterling RP, Pardanani A, Vannucchi AM. MIPSS70+ Version 2.0: Mutation and Karyotype-Enhanced International Prognostic Scoring System for Primary Myelofibrosis. J Clin Oncol. 2018 Jun 10;36(17):1769-1770. doi: 10.1200/JCO.2018.78.9867. Epub 2018 Apr 30. No abstract available. PMID 29708808
- [Background] Cervantes F. How I treat myelofibrosis. Blood. 2014 Oct 23;124(17):2635-42. doi: 10.1182/blood-2014-07-575373. Epub 2014 Sep 16. PMID 25232060
- [Background] Mesa RA. Ruxolitinib, a selective JAK1 and JAK2 inhibitor for the treatment of myeloproliferative neoplasms and psoriasis. IDrugs. 2010 Jun;13(6):394-403. PMID 20506062
- [Background] Heine A, Brossart P, Wolf D. Ruxolitinib is a potent immunosuppressive compound: is it time for anti-infective prophylaxis? Blood. 2013 Nov 28;122(23):3843-4. doi: 10.1182/blood-2013-10-531103. No abstract available. PMID 24288410